CLINICAL TRIAL: NCT01077180
Title: Rheos Feasibility Trial- A Study of Baroreflex Hypertension TherapyTM in Refractory Hypertension
Brief Title: Rheos Feasibility Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CVRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 360005-001
Record Dates: First submitted 2010-02-25; First posted 2010-02-26 (Estimated); Last update posted 2019-07-02 (Actual); Status verified 2016-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Rheos Device (Experimental)
  Interventions: Device: Implantation of the Rheos System
- Medical Management (Active Comparator)
  Interventions: Other: Standard of care medical management

INTERVENTIONS:
Device: Implantation of the Rheos System — Open label
  Arms: Rheos Device
Other: Standard of care medical management — Patients will continue with medical therapy for standard of care of their hypertension.
  Arms: Medical Management

SUMMARY:
The Rheos Feasibility Trial is designed to assess safety, device performance, and protocol parameters of the CVRx Rheos Baroreflex Therapy in patients with severe hypertension that are refractory to full drug therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 21 years of age.
2. Have been assessed to have bilateral carotid bifurcations located at or below C3-C4.
3. Have an office cuff systolic blood pressure greater than or equal to 160 mmHg and a 24-hour ambulatory systolic blood pressure greater than or equal to 150 mmHg despite at least one month of full therapy with at least three (3) anti-hypertensive medications, of which at least one (1) must be a diuretic.
4. Must be certified by the investigator hypertension specialist as compliant with taking full doses of medication.
5. Have signed a CVRx approved informed consent for participation in this study.

Exclusion Criteria:

1. Have been diagnosed with:

   * Baroreflex failure
   * Cardiac bradyarrhythmias
   * Chronic atrial fibrillation
2. Had a heart transplant
3. Have carotid atherosclerosis producing a 50% or greater reduction in linear diameter as determined by ultrasound or angiographic evaluation as determined within six months of enrollment in the trial.
4. Have Grade C ulcerative plaques in the carotid artery as determined by ultrasound or angiographic evaluation.
5. Have prior surgery or radiation in either carotid sinus region.
6. Currently have implanted electrical medical devices such as cardiac pacing, defibrillation or neurologic stimulation systems.
7. Are pregnant or contemplating pregnancy during the 13-month follow-up period.
8. Currently undergoing dialysis.
9. Have hypertension secondary to a treatable cause.
10. Have clinically significant cardiac valvular disease.
11. Are unable or unwilling to fulfill the protocol medication compliance and follow-up requirements.
12. Are unlikely to survive the protocol follow-up period.
13. Are enrolled in another concurrent clinical trial.

    -

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2005-01; Primary Completion 2007-12 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Rheos Feasibility Study | 13 months
  To summarize the efficacy of the Rheos System by estimating the reduction of systolic blood pressure associated with activation of the Rheos System at 4 and 13 months post implant when compared to baseline (1-month post implant).
  To describe the safety of the Rheos System by summarizing all system related adverse events and estimating the serious sytem related event-free rate through 4 and 13 months post-implant.